CLINICAL TRIAL: NCT04231578
Title: Couple HOPES: Initial Development of a Guided, Internet-delivered Couple Intervention for Posttraumatic Stress Disorder (PTSD) and Relationship Enhancement
Brief Title: Couple HOPES (Helping Overcome PTSD and Enhance Satisfaction)
Acronym: HOPES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Candice Monson, Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIHR-IRSC:0525007697; CIHR-IRSC:0525007697 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR) 2018-2019 Foundation Grant); W7714-207266 (Other Grant/Funding Number: National Defence Security Orders and Directives)
Record Dates: First submitted 2019-12-18; First posted 2020-01-18 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Self-help; Internet-delivered intervention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participating couples are either non-randomized in early phases of project or randomized to either immediately receive the Internet-delivered Couple HOPES intervention or to a delayed intervention group, where they receive access to Couple HOPES 8 weeks later.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Couple HOPES (Experimental): Immediately assigned to receive seven modules of an Internet-delivered self-help intervention with paraprofessional coaching for PTSD completed at the participant's own pace within 8 weeks.
  Interventions: Behavioral: Couple HOPES Guided, Internet-Delivered, Self-Help Intervention
- Delayed Intervention (No Intervention): Participants will not receive Couple HOPES for the first 8 weeks, and complete assessments at the beginning, middle, and end of this period. After this 8-week delay, participants will then receive seven modules of an Internet-delivered self-help intervention with paraprofessional coaching for PTSD completed at the participant's own pace within 8 weeks.

INTERVENTIONS:
Behavioral: Couple HOPES Guided, Internet-Delivered, Self-Help Intervention — Couple HOPES is a guided self-help intervention for individuals with PTSD and their partners based on Cognitive-Behavioral Conjoint Therapy for PTSD (Monson & Fredman, 2012). This intervention consists of text and video-based content across seven intervention modules and phone and online-based coaching sessions with a paraprofessional. Participants are able to complete these modules in their own home or private location of their choosing. The primary outcomes are PTSD symptoms, relationship satisfaction, and the mental health and wellbeing of partners of those with PTSD.
  Arms: Immediate Couple HOPES

SUMMARY:
Posttraumatic stress disorder (PTSD) is a common and disabling condition associated with intimate relationship problems and mental health problems in partners of those with PTSD. Recognizing the need to improve access to evidence-based interventions for those with PTSD and their families, our team has developed an Internet-delivered, self-help intervention to improve PTSD, enhance relationships, and improve partners' mental health: Couple HOPES (Helping Overcome PTSD and Enhance Satisfaction). Couple HOPES presents text and video-based content across seven self-help intervention modules, with modest support from paraprofessional coaches. Although the Couple HOPES platform has been developed, it remains uncertain whether Couple HOPES is feasible, usable, and efficacious in reducing PTSD and enhancing intimate relationship functioning. The proposed project aims to refine and finalize Couple HOPES with couples that include a veteran, service member or first responder with significant PTSD symptoms. This project includes initial testing of the intervention's preliminary efficacy, safety, and feasibility in a series of 10 couples (Phase 1), then in an uncontrolled trial of 20 couples (Phase 2), and then a randomized clinical trial comparing its efficacy to a delayed intervention control condition in 70 couples. Potential benefits of this study include couples learning new skills to reduce PTSD symptoms and enhance relationship functioning, although this is not guaranteed. Risks include participants finding the assessments distressing, or possible worsening of PTSD symptoms or relationship functioning. These risks will be mitigated by continuous monitoring of PTSD symptoms, relationship functioning, and adverse events, and intervention by study staff.

ELIGIBILITY:
Inclusion Criteria:

* Individual who is a Canadian military member, veteran, or first responder with clinically significant levels of PTSD symptoms
* Must be willing to be audio-recorded for coaching sessions
* Intimate partner willing to participant and complete intervention modules together
* Access to high speed internet

Exclusion Criteria:

* Elevated suicide risk
* Severe physical aggression between partners in the past year
* Clinically significant PTSD symptoms in both members of the dyad

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-5 (PCL-5) with change measured as mean change from baseline | Baseline, week 3, week 8, approximately once a week during treatment (for up to 8 weeks), after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
  Scores on the PCL-5 range from 0 to 80, with 80 being the most severe PTSD symptoms.
Couple Satisfaction Index (CSI-4) with change measured as mean change from baseline | Baseline, week 3, week 8, approximately once a week during treatment (for up to 8 weeks), after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
  Score on the CSI-4 range from 0 to 21, with 21 being the most satisfied.

SECONDARY OUTCOMES:
Mean change from baseline on Ineffective Arguing Inventory | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
  Score range from 0 to 40, with 40 representing highly ineffective arguing.

OTHER OUTCOMES:
Significant Others' Responses to Trauma Scale with change measured as mean change from baseline | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
  Scores range from 0 to 76, with 76 representing high partner accommodation.
Mean change from baseline on depression as measured by the Patient Health Questionnaire | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
  Scores range from 0 to 27, with 27 being the most depressed.
Mean change from baseline on alcohol use as measured by the Alcohol Use Disorders Identification Test: Self-Report Version | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
  Scores range from 0 to 40, with a higher score signifying an alcohol use disorder.
Mean change from baseline in drug use based on the Drug Abuse Screen Test | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
  Scores range from 0 to 10, with 10 being a severe level of problems related to drug abuse.
Generalized Anxiety Disorder symptoms with change measured as mean change from baseline | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
  Scores range from 0 to 21, with 21 representing the highest level of anxiety.
State-Trait Anger Expression Inventory with change measured as mean change from baseline | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
  Scores range from 0 to 40, with 40 representing higher levels of anger.
Mean change from baseline in perceived health measured with one item "How satisfied are you with your health" | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
  Scores range from 1 to 5, with 5 being the most satisfied.
Trauma-Related Guilt Inventory with change measured as mean change from baseline | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
Mean change from baseline in work functioning measured with one item "Please rate your ability to function at work. If you do not work outside the home, please rate your ability to complete household tasks." | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
Mean change from baseline in quality of life measured with one item "How would you rate your quality of life." | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
Participant ratings of intervention satisfaction as indicated by the Client Satisfaction Questionnaire | After 7 modules are completed or 8 weeks into treatment
Feasibility as measured by number of treatment sessions attended and rate of participant dropout | Once a week during treatment (for up to 8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Candice M Monson, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Candice M. Monson, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monson, C. M., & Fredman, S. J. (2012). Cognitive-behavioral conjoint therapy for PTSD: Harnessing the healing power of relationships. New York, NY: Guilford.
- [Derived] Fitzpatrick S, Crenshaw AO, Valela R, Samonas C, Earle EA, Goss S, Hernandez KM, Bushe J, Varma S, Proctor D, Wagner AC, Goenka K, Luxor O, Collins A, Morland L, Shields N, Roth M, Doss BD, Schumm J, Monson CM. A randomized controlled trial testing couple HOPES: An online, self-help couples' intervention for posttraumatic stress disorder. J Consult Clin Psychol. 2025 Aug;93(8):580-594. doi: 10.1037/ccp0000965. PMID 40811121
- [Derived] Crenshaw AO, Whitfield KM, Collins A, Valela R, Varma S, Landy MSH, Ip J, Donkin V, Earle E, Siegel A, Samonas C, Bushe J, Mensah DH, Xiang A, Doss BD, Morland L, Wagner AC, Fitzpatrick S, Monson CM. Partner outcomes from an uncontrolled trial of Couple HOPES: A guided online couple intervention for posttraumatic stress disorder and relationship enhancement. J Trauma Stress. 2023 Feb;36(1):230-238. doi: 10.1002/jts.22878. Epub 2022 Sep 18. PMID 36116104
- [Derived] Monson CM, Wagner AC, Crenshaw AO, Whitfield KM, Newnham CM, Valela R, Varma S, Di Bartolomeo AA, Fulham L, Collins A, Donkin V, Mensah DH, Landy MSH, Samonas C, Morland L, Doss BD, Fitzpatrick S. An uncontrolled trial of couple HOPES: A guided online couple intervention for PTSD and relationship enhancement. J Fam Psychol. 2022 Sep;36(6):1036-1042. doi: 10.1037/fam0000976. Epub 2022 Mar 10. PMID 35266773